CLINICAL TRIAL: NCT03927794
Title: Biomimetic Remineralization Using Self-Assembling Peptide P11-4 in the Prevention and Treatment of Early Carious Lesions in Primary Anterior Teeth: An In-Vivo and In-Vitro Study
Brief Title: Remineralization of White Spot Lesions Using Self-Assembling Peptide P11-4 in Primary Anterior Teeth A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nour Wahba, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED 19-1 D
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: White Spot Lesions [Initial Caries] on Smooth Surface of Tooth
Keywords: Self-Assembling Peptide P11-4; Biomimetic Remineralization; White spot lesions; Primary Anterior Teeth; Biomimetic Mineralization

STUDY DESIGN:
Intervention Model Description: 2 Groups where group A will receive self-assembling peptide P11-4 and group B will receive topical fluoride varnish.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded trial where patients won't know to which group they are assigned and where the outcome assessor will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Assembling Peptide P11-4 (Experimental): Twenty two teeth affected with white spot lesions of ICDAS II score 1-2 will be assessed at baseline using ICDAS II Scoring and Light Induced Fluorescence by Soprolife System.
  Then they will receive the intervention by the self-Assembling Peptide P11-4 at Day 0 and will be followed up at 3 months, 6 months and 1 year.
  Interventions: Other: Self-Assembling Peptide P11-4
- 5% Fluoride Varnish (Active Comparator): Twenty two teeth affected with white spot lesions of ICDAS II score 1-2 will be assessed as baseline using ICDAS II Scoring and Light Induced Fluorescence by Soprolife System.
  Then they will receive Topical Fluoride Varnish at Day 0 and will be followed up at 3 months, 6 months and 1 year.
  Interventions: Other: Self-Assembling Peptide P11-4

INTERVENTIONS:
Other: Self-Assembling Peptide P11-4 — Self-Assembling Peptide P11-4 promotes subsurface biomimetic remineralization of enamel. It is a small peptide comprising 11 amino acids that when applied to an initial carious lesion diffuses into the body of the lesion, re-assembles itself into fibrils forming larger fibers and hence a 3-dimensional (3-D) matrix is formed. Natural remineralization driven by saliva is promoted through the surface of the P11-4 by increasing the surface area for calcium phosphate deposition. As a result, mineralization of the subsurface lesion occurs possibly due to the formation of de novo hydroxyapatite crystals on the surface of the P11-4 fibers.
  Other Names: Curodont Repair

SUMMARY:
This study is a randomized controlled clinical trial on primary anterior teeth of 3-5 year-old patients suffering from white spot lesions (ICDAS system II scores 1-2).

Forty four teeth will be divided into two groups where Group 1 (n=22 teeth) will receive Self-Assembling Peptide P11-4.

Group 2 (n=22 teeth) will receive Topical Fluoride Varnish Application.

Assessment will be done at baseline using the International Caries Detection and Assessment System II (ICDAS II) scoring system and Light Induced Fluorescence using Soprolife System (Acteon, La Ciotat, France) and then after 3 months, 6 months and 1 year. The assessment of the baseline and follow up data will be performed by the main investigator.

DETAILED DESCRIPTION:
Patients aged 3-5 years with 44 teeth affected by white spot lesions (WSL) on their primary anterior teeth (ICDAS II scores 1-2) will be selected by simple random sample.

A minimum of 1 tooth and a maximum of 12 teeth affected by WSL in each patient can be included.

Subjects whose parents are willing and able to maintain good oral hygiene for their children and attend study visits.Subjects not on medication affecting their salivary flow and medically free (ASA class I).

1. All participating patients' parents will sign an informed consent.
2. Patients will receive oral information on oral health education on how to maintain a proper oral hygiene and proper diet consumption.
3. They will be given manual tooth brushes and non-fluoridated tooth pastes to use during the study. The tooth brushes will be replaced every 3 months and the tooth pastes will be replaced whenever they are empty.

5) Every patient will receive prophylaxis (polishing) using non-fluoridated prophylaxis paste prior to the commencement of treatment to avoid possible confounding factors.

6) Then each patient will be assigned to one of the two groups:

Group A: Self Assembling Peptides P11-4 (SAP Curodont Repair, Credentis, Windisch, Switzerland) 1) Twenty two teeth will receive treatment by self-assembling peptides P11-4 at baseline and will be followed up at 3 months, 6 months and 1 year using the above-mentioned measurements.

Group B: Topical Fluoride Varnish (Duraphat Varnish containing 22,600ppm fluoride, Colgate-Palmolive, USA)

1) Twenty two teeth will receive treatment by topical fluoride varnish at Day 0 and will be followed up after 3 months, 6 months and 1 year using the above-mentioned measurements.

The assessment of the baseline and follow up data will be performed by the main investigator.

Assessment will be done at baseline using the ICDAS II and Light Induced Fluorescence using Soprolife System (Acteon, La Ciotat, France) and then at 3 months, 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients ASA Class I.
* ≥1 Primary Anterior Teeth with early carious lesions of ICDAS scores 1-2.
* Subjects whose parents are willing and able to maintain good oral hygiene for their children and attend study visits.
* Patients aged between 3-5 years.
* Subjects with a minimum of 1 and a maximum of 12 primary anterior teeth with early carious lesions of ICDAS II scores 1-2.

Exclusion Criteria:

* Primary anterior teeth in which carious lesions are scored with ICDAS ≥3.
* Subjects on medication that affects the salivary flow rate.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Remineralization of white spot lesions | One year
  Remineralizing efficacy of self-assembling peptide P11-4 versus fluoride varnish using light induced fluorescence (Soprolife Camera). Patients' white spot lesions will be examined using Soprolife camera to identify the demineralized areas. At 3 months, 6 months, and 1 year after treatment their lesions will be re-assessed and compared with baseline data.

SECONDARY OUTCOMES:
Caries progression or regression by ICDAS II system | One year
  Caries progression/ regression using ICDAS II system. If the score has increased to ICDAS 3 or more indicates caries progression and if it decreases to 0-1 this indicates caries regression; if score remains the same this indicates no change in lesion.
  Each lesion will be scored at baseline by ICDAS II system and then at 3 months, 6 months, and 1 year.
- Patient satisfaction/dissatisfaction | 1 day
  - Patient satisfaction/dissatisfaction regarding each intervention using a Caregiver Satisfaction Questionnaire for each patient undergoing the treatment. This will be done on the same visit of treatment after its application.

CONTACTS AND LOCATIONS:
Overall Officials: Noha SA Kabil, PHD, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alkilzy M, Santamaria RM, Schmoeckel J, Splieth CH. Treatment of Carious Lesions Using Self-Assembling Peptides. Adv Dent Res. 2018 Feb;29(1):42-47. doi: 10.1177/0022034517737025. PMID 29355413
- [Result] Alkilzy M, Tarabaih A, Santamaria RM, Splieth CH. Self-assembling Peptide P11-4 and Fluoride for Regenerating Enamel. J Dent Res. 2018 Feb;97(2):148-154. doi: 10.1177/0022034517730531. Epub 2017 Sep 11. PMID 28892645
- [Result] Kind L, Stevanovic S, Wuttig S, Wimberger S, Hofer J, Muller B, Pieles U. Biomimetic Remineralization of Carious Lesions by Self-Assembling Peptide. J Dent Res. 2017 Jul;96(7):790-797. doi: 10.1177/0022034517698419. Epub 2017 Mar 27. PMID 28346861
- [Result] Silvertown JD, Wong BPY, Sivagurunathan KS, Abrams SH, Kirkham J, Amaechi BT. Remineralization of natural early caries lesions in vitro by P11 -4 monitored with photothermal radiometry and luminescence. J Investig Clin Dent. 2017 Nov;8(4). doi: 10.1111/jicd.12257. Epub 2017 Jan 4. PMID 28052551